CLINICAL TRIAL: NCT00004338
Title: Study of Zinc for Wilson Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Michigan (Other)
Purpose: Treatment
Other Study IDs: 199/11897; UMMC-310
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Wilson Disease
Keywords: Wilson disease; inborn errors of metabolism; rare disease
MeSH Terms: conditions — Hepatolenticular Degeneration; Metabolism, Inborn Errors; Rare Diseases | interventions — Zinc Acetate

INTERVENTIONS:
Drug: zinc acetate

SUMMARY:
OBJECTIVES: I. Establish the safety and efficacy of extended maintenance zinc therapy in 200 patients with Wilson disease.

II. Establish further the role of zinc in the prophylactic treatment of presymptomatic patients by increasing the current cohort from 80 to at least 100 patients.

III. Establish further the role of zinc therapy in pregnant patients with Wilson disease.

IV. Establish further the role of zinc therapy in children with Wilson disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients receive copper regulation therapy with zinc acetate: an existing cohort on maintenance therapy will be followed for long-term data collection; presymptomatic patients are treated prophylactically; and pregnant patients are evaluated for fetal outcome. All patients are evaluated for copper balance, clinical control, and toxicity.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA: Wilson disease Presymptomatic, pregnant, and children 16 years or younger patients eligible Patient age: Any age, including children

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 1993-10

CONTACTS AND LOCATIONS:
Overall Officials: George J. Brewer, Study Chair — University of Michigan
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Brewer GJ, Yuzbasiyan-Gurkan V, Johnson V. Treatment of Wilson's disease with zinc. IX: Response of serum lipids. J Lab Clin Med. 1991 Nov;118(5):466-70. PMID 1940587
- [Background] Yuzbasiyan-Gurkan V, Grider A, Nostrant T, Cousins RJ, Brewer GJ. Treatment of Wilson's disease with zinc: X. Intestinal metallothionein induction. J Lab Clin Med. 1992 Sep;120(3):380-6. PMID 1517684
- [Background] Brewer GJ, Yuzbasiyan-Gurkan V, Johnson V, Dick RD, Wang Y. Treatment of Wilson's disease with zinc XII: dose regimen requirements. Am J Med Sci. 1993 Apr;305(4):199-202. doi: 10.1097/00000441-199304000-00001. PMID 8475943
- [Background] Brewer GJ, Yuzbasiyan-Gurkan V, Johnson V, Dick RD, Wang Y. Treatment of Wilson's disease with zinc: XI. Interaction with other anticopper agents. J Am Coll Nutr. 1993 Feb;12(1):26-30. doi: 10.1080/07315724.1993.10718278. PMID 8440814
- [Background] Brewer GJ, Dick RD, Yuzbasiyan-Gurkan V, Johnson V, Wang Y. Treatment of Wilson's disease with zinc. XIII: Therapy with zinc in presymptomatic patients from the time of diagnosis. J Lab Clin Med. 1994 Jun;123(6):849-58. PMID 8201263
- [Background] Brewer GJ, Johnson V, Kaplan J. Treatment of Wilson's disease with zinc: XIV. Studies of the effect of zinc on lymphocyte function. J Lab Clin Med. 1997 Jun;129(6):649-52. doi: 10.1016/s0022-2143(97)90200-6. PMID 9178732
- [Background] Beck FW, Prasad AS, Kaplan J, Fitzgerald JT, Brewer GJ. Changes in cytokine production and T cell subpopulations in experimentally induced zinc-deficient humans. Am J Physiol. 1997 Jun;272(6 Pt 1):E1002-7. doi: 10.1152/ajpendo.1997.272.6.E1002. PMID 9227444